CLINICAL TRIAL: NCT01497691
Title: A Randomized Controlled Trial of Noninvasive Positive Airway Pressure in the Pediatric Emergency Department for the Treatment of Acute Asthma Exacerbations
Brief Title: Noninvasive Positive Airway Pressure in the Pediatric Emergency Department for the Treatment of Acute Asthma Exacerbations
Acronym: RCT BiPAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit participants
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111491
Record Dates: First submitted 2011-12-16; First posted 2011-12-22 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Asthma; Pediatrics; BiPAP; Noninvasive Positive Pressure Ventilation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Other): This group will receive all standard of care therapies as per the pediatric ED Asthma Severity Protocol.
  Interventions: Device: USCOM
- Sham NIPPV (Sham Comparator): This group will receive all standard of care therapies as per the pediatric ED Asthma Severity Protocol. All nebulized treatments will be given via the NIPPV/BiPAP machine. The pressure settings will be fixed at a positive end-expiratory pressure (PEEP) of 5-8 cm H2O.
  Interventions: Device: NIPPV (PALMtop PTV); Device: Volumetric CO2 (NM3); Device: USCOM
- BiPAP (Active Comparator): This group will receive all standard of care therapies as per the pediatric ED Asthma Severity Protocol. All nebulized treatments will be given via the NIPPV/BiPAP machine. Settings will be adjusted based on the age and clinical presentation of the child.
  Interventions: Device: NIPPV (PALMtop PTV); Device: Volumetric CO2 (NM3); Device: USCOM

INTERVENTIONS:
Device: NIPPV (PALMtop PTV) — PALMtop PTV Models 8/10 aka CareFusion EnVe The primary study device is the PALMtop PTV. It is the NIPPV/BiPAP device used in this study. It is FDA approved for use in children who weigh 5 kilograms or greater (#K070594).
  Arms: BiPAP; Sham NIPPV
Device: Volumetric CO2 (NM3) — The NM3 is FDA approved (#K091459) for spirometric and carbon dioxide monitoring as well as continuous, non-invasive monitoring of arterial oxygen saturations and pulse rates in neonatal and pediatric patients in the emergency department.
  Arms: BiPAP; Sham NIPPV
Device: USCOM — The USCOM a non-invasive ultrasonic device that is FDA approved for monitor beat-to-beat cardiac hemodynamics in adult and pediatric patients (#K043139). It will be used in an attempt to better understand the underlying physiology of NIPPV use.

SUMMARY:
Previous investigations and anecdotal experience have shown safety and utility of Noninvasive Positive Pressure Ventilation/Bilevel Positive Airway Pressure (NIPPV/BiPAP) for the treatment of asthma in children. If NIPPV/BiPAP can be shown to have a beneficial effect in children with respiratory insufficiency, emergency department and ICU stays may be shortened, and the need for more invasive and dangerous airway procedures may be decreased. This would result in a change in the standard of care for asthma treatment in emergency departments. The investigators hypothesis is that the use of this new NIPPV, in conjunction with current standard of care therapies, in acute moderate to severe asthma exacerbations will lead to a more rapid improvement in patient ventilation, faster resolution of respiratory distress, and overall improved secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years old
* For subjects 3 years and older, a known history of asthma as diagnosed by the PCP or per the Vanderbilt problem list
* For children ages 2-3 years, four or more episodes of wheezing in the past year that lasted more than 1 day and affected sleep AND one of the following: parental history of asthma, a physician diagnosis of atopic dermatitis, or evidence of sensitization to aeroallergens
* Acute asthma exacerbation
* Pediatric Asthma Score (PAS) ≥ 8
* Parents willing and able to sign consent
* Children over the age of 6 willing to provide assent

Exclusion Criteria:

* History of congenital heart disease, chronic respiratory disease including bronchopulmonary dysplasia, cystic fibrosis, pulmonary hypertension or any chronic lung disease other than asthma
* History of sickle cell disease
* Recently diagnosed pneumonia
* Current tracheostomy, on home ventilator or home oxygen requirement
* Recent diabetic ketoacidosis
* Requiring immediate intubation
* Weight less than 5 kilograms
* Any contraindication to BiPAP use including altered mental status, recent bowel surgery, intractable vomiting, inability to protect airway
* A history of prematurity of ≤ 30 weeks gestation

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Estimated); Primary Completion 2013-11-19 (Actual); Study Completion 2013-11-19 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Asthma Score | Every 30 minutes while the subject is enrolled
  The primary outcome indicator will be a decrease in PAS to ≤ to 7 to occur 3 hours faster in the NIPPV/BiPAP group as compared to the control group (median expected time to PAS 7 ≤ in BiPAP group is 5 hours; median expected time to PAS ≤ 7 in control group is 8 hours; hazard ratio is 1.6). A total sample size of 366 (122 in each group) is required for 80% power and a significance level of 0.05 (2 tailed test). With an estimated 20% drop out rate will anticipate 147 subjects enrolled per arm for a total of 441 subjects enrolled.

SECONDARY OUTCOMES:
Volumetric end tidal CO2 trend | Continuous while the subject is enrolled
  Measurement of volumetric end tidal CO2 trend with the NICO2® Respiratory volumetric capnography CO2 monitors
Respiratory parameters | Continuous while the subject is enrolled
  Analysis of flow loops captured by the NIPPV device, the delta pediatric asthma scores at each time point and changes in individual pulmonary parameters (respiratory rate, oxygen requirement, oxygen saturation).
Cardiac output | Continuous while the subject is enrolled
  Changes in cardiac parameters as measured by the USCOM
Intubation and complication rates | Continuous observation
  Documentation of intubation rate and possible complications including but not limited to hypotension, vomiting, agitation, skin irritation, pneumothorax, barotrauma effects and death.
Length of hospital stay | Retrospectively upon completion of study
  Decrease length of hospital stay if placed on NIPPV. This will include looking at the disposition of the subject from the pediatric emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Abby M Williams, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States